CLINICAL TRIAL: NCT05492045
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 Combination Therapy in Subjects With KRAS G12C-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate D-1553 in Combination Therapy in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adjustment of drug development strategy.
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1553-105
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1b Dose escalation of D-1553 combination therapies (Experimental): Phase 1b will determine maximal tolerated dose and/or recommended phase 2 dose of D-1553 in combination with immunotherapy or targeted therapy in patients with KRAS G12C-mutated locally advanced or metastatic NSCLC.
  Interventions: Drug: D-1553; Drug: Other
- Phase 2 of D-1553 combination therapies (Experimental): Phase 2 will evaluate the efficacy and safety of D-1553 combined with immunotherapy or targeted therapy in patients with KRAS G12C-mutated locally advanced or metastatic NSCLC.
  Interventions: Drug: D-1553; Drug: Other

INTERVENTIONS:
Drug: D-1553 — D-1553 is a novel, targeted KRasG12C inhibitor that is being developed as a potential oral agent for advanced or metastatic solid tumors with KRasG12C mutation.
Drug: Other — Standard treatment of NSCLC.

SUMMARY:
This is a Phase 1b/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 Combination Therapy in Subjects with KRAS G12C-mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject with histologically proven, locally advanced or metastatic NSCLC for which has no standard treatment or the subject has been previously treated with first- or second-line systemic therapy.
* Subject has KRasG12C mutation in tumor tissue or other biospecimens containing cancer cells or DNA. Historical, local laboratory result (up to 5 years prior to this study) can be used for Phase 1 subjects. Phase 2 subjects must be tested for KRasG12C mutation by a local laboratory.
* Subject has measurable disease according to RECIST v1.1. For phase 1b subjects who have no measurable lesions but whose disease can be evaluated are also acceptable.

Exclusion Criteria:

* Subject with unstable or progressive central nervous system (CNS) metastases.
* Subjects with clinically significant cardiovascular disease.
* Subject with interstitial lung disease (ILD) or any active systemic infection including but not limited to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Subject has impaired gastrointestinal (GI) function or GI diseases that may significantly alter the absorption or metabolism of oral medications.
* Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Subject incidence of Dose-limiting toxicities (DLT) | Through out the DLT period, approximately 21 days
  Subject incidence of Dose-limiting toxicities (DLT)
Number of subjects participants with adverse events | Till study completion, approximately 3 years
  Number of subjects participants with adverse events
Antitumor activity of D-1553 in subjects with advanced or metastatic NSCLC with KRASG12C mutation | Till study completion, approximately 3 years
  Overall Response Rate (ORR, Complete Response [CR] + Partial Response [PR])

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Cancer Hospital of the University of Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No